CLINICAL TRIAL: NCT02076594
Title: A Randomized Phase III Study Of Low-Docetaxel Oxaliplatin, Capecitabine (Low-Tox) Vs Epirubicin, Oxaliplatin And Capecitabine (Eox) In Patients With Locally Advanced Unresectable Or Metastatic Gastric Cancer
Brief Title: Low-Tox Vs Eox In Patients With Locally Advanced Unresectable Or Metastatic Gastric Cancer
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The interim analysis performed on 09 November 2018, showed the failure to achieve the primary objective of effectiveness of the experimental treatment.
Sponsor: Gruppo Italiano per lo studio dei Carcinomi dell'Apparato Digerente (Other)
Collaborators: Regione Lombardia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LEGA; 2011-005537-39 (EudraCT Number)
Record Dates: First submitted 2013-08-20; First posted 2014-03-03 (Estimated); Last update posted 2019-10-09 (Actual); Status verified 2019-01

CONDITIONS: Locally Advanced Unresectable Gastric Cancer; Metastatic Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Docetaxel; Epirubicin; Oxaliplatin; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Docetaxel & Oxaliplatin & Capecitabine (Experimental): Patients will receive cycles every 3 weeks of Docetaxel (35 mg/ m2, intravenous at days 1 and 8 by 1-hour infusion)and Oxaliplatin (80 mg/ m2, intravenous at day 1 by 2-hour infusion) and Capecitabine (750 mg/ m2, oral tablets of 500 and 150 mg, x2 daily for 2 weeks)
  Interventions: Drug: Docetaxel; Drug: Oxaliplatin; Drug: Capecitabine
- Epirubicin & Oxaliplatin & Capecitabine (Experimental): Patients will receive cycles every 3 weeks of Epirubicin (50 mg/ m2, intravenous on day 1 by 2-hour infusion)and Oxaliplatin (130 mg/ m2, intravenous on day 1 by 2-hour infusion) and Capecitabine (625 mg/ m2,oral tablets of 500 and 150 mg, x2 daily for 3 weeks)
  Interventions: Drug: Epirubicin; Drug: Oxaliplatin; Drug: Capecitabine

INTERVENTIONS:
Drug: Docetaxel — Powder for solution for infusion
  Other Names: Taxotere 20 mg/mL
  Arms: Docetaxel & Oxaliplatin & Capecitabine
Drug: Epirubicin — Solution for infusion
  Other Names: Farmorubicina 2mg/mL
  Arms: Epirubicin & Oxaliplatin & Capecitabine
Drug: Oxaliplatin — Powder for solution for infusion
  Other Names: Eloxatin 5 mg/mL
Drug: Capecitabine — Film coated tablets
  Other Names: Xeloda 150 mg; Xeloda 500 mg

SUMMARY:
This is a randomized, parallel group, non-blinded phase III trial. Patients with advanced (locoregional or metastatic) gastric cancer not previously treated with chemotherapy for this stage will be randomized in a 1:1 ratio to receive low-TOX (arm A) or EOX (arm B). Randomization will be stratified by performance status (ECOG 0, 1 and 2).

DETAILED DESCRIPTION:
Although the incidence of the adenocarcinoma of the stomach is slowly decreasing, gastric cancer represents the second worldwide cause of cancer death after lung cancer. In patients with advanced disease, chemotherapy improves survival and quality of life. Combinations of two or three drugs including a platin derivative (cisplatin or oxaliplatin), a fluoropyrimidine (5FU or capecitabine) and an anthracycline (usually epirubicin) have demonstrated superiority compared to single or double agent therapy and are the current standard. As of today there are no published studies comparing anthracycline-based to taxane-based three-drug regimens. The objective of the present study is to compare EOX as evaluated in REAL-2 to the low-TOX regimen consisting of docetaxel, oxaliplatin and capecitabine. Low-TOX is expected to be better tolerated than the original DCF regimen. The study will be performed in the HER2 negative patients.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent prior to beginning protocol specific procedures
* Male or female > 18 years of age
* Histologically proven diagnosis of adenocarcinoma of the stomach
* HER2 negative tumor or HER2+ tumors not qualifying for herceptin therapy
* Locally advanced (non resectable) or metastatic gastric cancer
* Presence of measurable disease with at least one measurable lesion by means of CT scan or MRI in not previously irradiated area(s) (according to RECIST criteria (version 1.1)
* Life expectancy of >/= 3 months
* ECOG performance status of 0-2 at study entry
* Neutrophils >/= 2.0 x 1000000000/L, platelets >/= 100 x 1000000000/L, and hemoglobin >/= 10 g/dL
* Bilirubin level either normal or </= 1.5 x ULN
* AST and ALT </= 2.5 X UNL (</= 5 x ULN if liver metastasis are present
* Alkaline phosphatase (ALP) </= 2.5 X ULN; patients with alkaline phosphatase > 2.5x ULN and AST and ALT </= 1.5 x ULN are equally eligible
* Serum creatinine < 1.5 x ULN. In presence border-line values, the calculated creatinine clearance should be >/= 60 mL/min
* Negative pregnancy test (if female in reproductive years)
* Effective contraception prior to study entry and for the duration of the study participation, for both male and female patients of child producing potential
* Able and willing to comply with scheduled visits, therapy plans and laboratory tests required in this protocol

Exclusion Criteria:

* Previous chemotherapy, except adjuvant treatment administered at least 1 year before study entry
* Concurrent chronic systemic immune therapy
* Any investigational agent(s) 4 weeks prior to entry
* Clinically relevant coronary artery disease or a history of a myocardial infarction or a history of hypertension not controlled by therapy within the last 12 months
* Known hypersensitivity to study drugs. Known grade 3 or 4 allergic reaction to any of the components of the treatment
* Known drug abuse/ alcohol abuse
* Acute or subacute intestinal occlusion and any other significant chronic gastrointestinal disease that might interfere with absorption of oral treatment
* History of clinically relevant psychiatric disability precluding informed consent
* Presence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule
* Pregnant or breastfeeding women
* Active uncontrolled infection(s)
* Positive for HIV serology and/or viral hepatitis B or C
* Any concurrent malignancy other than non-melanoma skin cancer, or carcinoma in situ of the cervix. (Patients with a previous malignancy but without evidence of disease for ≥ 5 years will be allowed to enter the trial)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 171 (Actual)
Dates: Start 2013-01; Primary Completion 2018-12 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | Measured as the time from randomization to the date of local or regional progression, distant metastasis, second primary malignancy or death, assessed up to 18 months of follow up
  To determine the progression free survival (PFS) of patients with locally advanced unresectable or metastatic gastric cancer treated with Docetaxel plus Oxaliplatin plus Capecitabine (Arm A) or with Epirubicin plus Oxaliplatin plus Capecitabine (Arm B)

SECONDARY OUTCOMES:
Overall Survival (OS) | Measured as the time from randomization to the date of death from any cause, assessed up to 18 months of follow up
  To assess overall survival (OS) of patients with locally advanced unresectable or metastatic gastric cancer treated with Docetaxel plus Oxaliplatin plus Capecitabine (Arm A) or with Epirubicin plus Oxaliplatin plus Capecitabine (Arm B)
Objective Response Rate (CR + PR) according to RECIST 1.1 guideline | Measured as the time from randomization, assessed up to 18 months of follow up
  To assess objective response rate (CR+PR)of patients with locally advanced unresectable or metastatic gastric cancer treated with Docetaxel plus Oxaliplatin plus Capecitabine (Arm A) or with Epirubicin plus Oxaliplatin plus Capecitabine (Arm B)
Disease control rate: CR + PR + SD lasting > 12 weeks | Measured as the time from randomization, assessed up to 18 months of follow up
  To assess disease control rate of patients with locally advanced unresectable or metastatic gastric cancer treated with Docetaxel plus Oxaliplatin plus Capecitabine (Arm A) or with Epirubicin plus Oxaliplatin plus Capecitabine (Arm B)
Tolerability of the treatments evaluated in term of occurrence of: side effects graded according to the NCI-CTCAE scale (version 4.0); serious adverse reactions, expected and unexpected | Measured as the time from randomization, assessed up to 18 months of follow up
  To assess tolerability of the treatments of patients with locally advanced unresectable or metastatic gastric cancer treated with Docetaxel plus Oxaliplatin plus Capecitabine (Arm A) or with Epirubicin plus Oxaliplatin plus Capecitabine (Arm B)

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Labianca, MD, Study Director — A.O. Papa Giovanni XXIII di Bergamo, Oncologia Medica; Enrico Cortesi, MD, Principal Investigator — Policlinico Umbero I di Roma, UOC Oncologia Medica B; Domenico Cristiano Corsi, MD, Principal Investigator — Ospedale Fatebenefratelli di Roma, Oncologia; Pietro Sozzi, MD, Principal Investigator — Ospedale degli Infermi di Biella, Oncologia; Luigi Cavanna, MD, Principal Investigator — AUSL di Piacenza, Oncologia Medica; Domenico Bilancia, MD, Principal Investigator — A.O. Ospedale San Carlo di Potenza, Oncologia Medica; Rosa Rita Silva, MD, Principal Investigator — ASUR Zona 6 di Fabriano, Oncologia; Nicola Fazio, MD, Principal Investigator — IRCCS Istituto Europeo di Oncologia di Milano, Tumori digestivi superiori e Neuroendocrini; Monica Giordano, MD, Principal Investigator — A. O. Sant'Anna di Como, Oncologia; Alessandro Bertolini, MD, Principal Investigator — Ospedale Civile di Sondrio, Oncologia Medica; Giovanni Ucci, MD, Principal Investigator — A.O. Ospedale Maggiore di Lodi, Oncologia; Donato Natale, MD, Principal Investigator — A.O. di Pescara - Oncologia; Daris Ferrari, MD, Principal Investigator — A.O. San Paolo di Milano, Oncologia Medica; Graziella Pinotti, MD, Principal Investigator — Ospedale di Circolo e Fondazione Macchi di Varese, Oncologia; Ermanno Rondini, MD, Principal Investigator — Ospedale di S. Maria Nuova di Reggio Emilia, Oncologia Medica; Massimo Cirillo, MD, Principal Investigator — Ospedale Sacro Cuore Don Calabria di Negrar, Oncologia Medica; Rosario Vincenzo Iaffaioli, MD, Principal Investigator — IRCCS Istituto Nazionale Tumori Fondazione Pascale di Napoli, Oncologia Medica Addominale; Andrea Ciarlo, MD, Principal Investigator — Ospedale Misericordia e Dolce di Prato, Oncologia Medica; Elena Piazza, MD, Principal Investigator — Ospedale L. Sacco di Milano, Oncologia; Libero Ciuffreda, MD, Principal Investigator — Azienda Ospedaliera Città della Salute e della Scienza di Torino, Oncologia Medica; Stefania Dell'Oro, MD, Principal Investigator — Ospedale di Circolo A. Manzoni di Lecco, Oncologia Medica; Fabrizio Artioli, MD, Principal Investigator — Ospedale di Carpi, Medicina Oncologica; Claudio Verusio, MD, Principal Investigator — Ospedale Generale Provinciale di Saronno, Oncologia Medica; Vincenzo Catalano, MD, Principal Investigator — A.O. Ospedali Riuniti Marche Nord - Presidio S. Salvatore Muraglia, Oncologia; Claudio Graiff, MD, Principal Investigator — ASDAA Bolzano, Oncologia Medica; Domenico Amoroso, MD, Principal Investigator — A.O. Ospedale Versilia di Camaiore, Oncologia Medica; Maria Di Bartolomeo, MD, Principal Investigator — Fondazione IRCCS Istituto Nazionale dei Tumori di Milano, Medicina Oncologica 1; Nicola Silvestris, MD, Principal Investigator — Istituto Tumori di Bari, Oncologia Medica; Maria C. Zavettieri, MD, Principal Investigator — OSPED. DI CIRCOLO SERBELLONI-GORGONZOLA - GORGONZOLA (MI); Enzo Veltri, MD, Principal Investigator — OSPEDALE SANTA MARIA GORETTI LATINA; Francesco Ferraù, MD, Principal Investigator — P.O. "SAN VINCENZO" TAORMINA - TAORMINA (ME); Giampaolo Tortora, MD, Principal Investigator — OSPEDALE POLICLINICO G.B. ROSSI (BORGO ROMA) DI VERONA; Sandro Barni, MD, Principal Investigator — A.O. TREVIGLIO-CARAVAGGIO - TREVIGLIO (BG); Mario Scartozzi, MD, Principal Investigator — A.O.U. di Cagliari - Presidio di Monserrato
Locations (25):
- Italy (25):
  - Istituto Tumori, Bari, BA
  - Azienda Ospedaliera Papa Giovanni XXIII, Bergamo, BG
  - A.O. Treviglio-Caravaggio, Treviglio, BG
  - Azienda Ospedaliera Universitaria di Cagliari, Monserrato, CA
  - Azienda Ospedaliera Sant'Anna, Como, CO
  - Ospedale di Circolo A. Manzoni, Lecco, LC
  - Ospedale Santa Maria Goretti Latina, Latina, LT
  - A.O. Ospedale Versilia, Camaiore, LU
  - P.O. "San Vincenzo" Taormina, Taormina, ME
  - Osped. Di Circolo Serbelloni-Gorgonzola, Gorgonzola, MI
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan, MI
  - IRCCS Istituto Europeo di Oncologia (IEO), Milan, MI
  - Azienda Ospedaliera San Paolo, Milan, MI
  - Ospedale L. Sacco, Milan, MI
  - Ospedale di Carpi, Carpi, MO
  - AUSL di Piacenza, Piacenza, PC
  - A.O. Ospedali Riuniti Marche Nord - Presidio S. Salvatore Muraglia, Pesaro, PE
  - A. O. di Pescara - Ospedale Civile Spirito Santo, Pescara, PE
  - Ospedale Misericordia e Dolce, Prato, PO
  - Azienda Ospedaliera Ospedale San Carlo, Potenza, PZ
  - Ospedale di S. Maria Nuova, Reggio Emilia, RE
  - Ospedale Fatebenefratelli, Roma, RM
  - Ospedale di Circolo e Fondazione Macchi di Varese, Varese, VA
  - Ospedale Sacro Cuore Don Calabria di Negrar, Negrar, VR
  - IRCCS Istituto Nazionale Tumori Fondazione Pascale, Napoli